CLINICAL TRIAL: NCT05034562
Title: Gallium-68 PSMA-11 PET in Participants With Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Per PI no participants enrolled
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-1203; NCI-2020-03699 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1203 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-06-10; First posted 2021-09-05 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Prostate Carcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (gallium Ga 68-labeled PSMA-11, PET/CT, PET/MRI) (Experimental): Patients receive gallium Ga 68-labeled PSMA-11 IV. 50-100 minutes after injection, patients then undergo a PET/CT scan or PET/MRI scan over 60 minutes.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68-labeled PSMA-11; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Gallium Ga 68-labeled PSMA-11 — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; Gallium Ga 68 PSMA-11; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT or PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase II trial studies how well gallium-68 PSMA-11 PET/CT or PET/MRI works in finding prostate cancer cells that have come back (recurrent) in patients with prostate cancer. Gallium-68 PSMA-11 is a type of radioactive compound, called a radiotracer, which is injected in the vein and can accumulate in tumor cells to generate a signal detected by PET/CT or PET/MRI imaging. This may help researchers in finding recurrent prostate cancer cells in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the positive predictive value (PPV) of gallium Ga 68-labeled PSMA-11 (68Ga-PSMA11) positron emission tomography/computed tomography (PET/CT) and positron emission tomography/magnetic resonance imaging (PET/MRI) on a patient level using histopathology or confirmatory imaging as a standard of truth (SoT).

SECONDARY OBJECTIVES:

I. To assess the PPV per-patient for 68Ga-PSMA-11 PET/CT and PET/MRI detection of tumor location confirmed by histopathology/biopsy alone.

II. Demonstrate the safety of 68Ga-PSMA-11 PET/CT or PET/MRI imaging in participants with prostate cancer.

III. Demonstrate the efficacy of 68Ga-PSMA-11 PET/CT or PET/MRI imaging to monitor response to treatment in participants with prostate cancer.

OUTLINE:

Patients receive gallium 68Ga-PSMA-11 intravenously (IV). 50-100 minutes after injection, patients then undergo a PET/CT scan or PET/MRI scan over 60 minutes.

After completion of study, patients are followed up at 30 and 90 days, then between 3-36 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven prostate cancer
* Rising prostate-specific antigen (PSA) after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy)
* Karnofsky performance status (KPS) >= 50 (Eastern Cooperative Oncology Group [ECOG]/World Health Organization [WHO] 0, 1, or 2)
* Ability to understand and willingness to provide informed consent
* Participants with known metastatic prostate cancer planned to undergo active systemic treatment

Exclusion Criteria:

* Unable to lie flat, still, or tolerate a PET or MRI scan
* Contraindication to optional furosemide administration including prior allergy or adverse reaction to furosemide or sulfa drugs. This exclusion criteria can be removed if furosemide is omitted as part of the PET imaging protocol if a second-generation scatter correction - (defined as either Ga-68 specific prompt gamma correction or multiple scatter model) is available for the used PET device

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Positive predictive value of 68Ga-PSMA-11 (gallium Ga 68-labeled PSMA-11) positron emission tomography (PET) | Up to 36 months
  Positive predictive value will be defined as true positive/(true positive + false positive). Positive predictive value on a per-participant and per-region-basis of 68Ga-PSMA-11 PET for detection of tumor location confirmed by histopathology/biopsy, clinical and conventional imaging follow-up will be calculated and reported along with the corresponding two-sided 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Ravizzini, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org